CLINICAL TRIAL: NCT00268619
Title: A Placebo-controlled, Double-blind, Randomized, Multicenter Study of Ramipril 5 and 10 mg Capsules and Insulin Infusion in Subjects With Unstable Coronary Syndromes
Brief Title: FOCUS:Focus On Coronary Unstable Syndromes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HOE498_3501
Record Dates: First submitted 2005-12-21; First posted 2005-12-22 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia | interventions — Ramipril

INTERVENTIONS:
Drug: Ramipril

SUMMARY:
Study objectives:

* To demonstrate that the acute administration of ramipril will control the inflammation process in patients with high-risk Acute Coronary Syndrome (ACS) as assessed by the high sensitivity C-reactive protein blood levels.
* To demonstrate that the normalization of blood glucose levels with intravenous insulin will improve the inflammation process during the acute phase of an ACS as assessed by Tumor necrosis factor alpha blood levels.

ELIGIBILITY:
Inclusion Criteria:

* Subject either not of childbearing potential or is not pregnant and agrees to use contraceptive measure for the duration of the study
* Subjects presenting within 12 hours after the last episode of chest pain with:

  * An accelerating pattern of anginal pain
  * A prolonged or recurrent anginal pain at rest or with minimal effort AND
  * Evidence of myocardial ischemia on ECG manifested by at least one of the following ECG criteria: - new persistent or transient ST-segment depression OR transient or reversible ST-segment elevation or new persistent or transient T-wave inversion OR Abnormal cardiac markers defined as: CK-MB greater than the upper limit of normal Troponin T or I level greater than the upper limit of normal.

Exclusion Criteria:

* Known or suspected pregnancy or actively breast-feeding
* Female of childbearing potential not using or planning to use a reliable method of contraception
* Treatment with Hormone Replacement Therapy at time of randomization
* Angina precipitated by obvious provoking factors
* Heart Failure defined as known ejection fraction less or equal to 40% or NYHA (New York Heart Association) class III pr IV
* Type I Diabetes Mellitus
* Type II diabetes requiring insulin therapy
* Hyperkaliemia
* Acute chronic inflammatory, collagen tissue disease, auto-immune disease or cancer and/or requiring the use of anti-inflammatory or anti-neoplastic agents at the time of randomization
* Use of a non-steriodal anti-inflammatory agent, coxibs, or anti-neoplasic agent within last 7 days
* Use of any oral or intra-venous steroidal agent in the last 7 days before study entry
* Uncontrolled hypertension
* Systolic pressure < 100 mmHg at randomization
* Likelihood of requiring treatment during the study period with drugs not permitted by the protocol
* Treatment with any investigational product or device in the last 4 weeks
* Previous participation into the trial
* History of hypersensitivity, allergy, or intolerance to Angiotensin-Converting Enzyme inhibitors.
* Severe cardiovascular diseases requiring urgent therapy
* Severe or co-morbid condition
* History of cancer not known to be disease free, with the exception of basal cell carcinoma of the skin
* Clinically important systemic disorder
* Impaired hepatic function
* Clinically important chronic or acute renal failure
* History of drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-06; Primary Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
To assess the highly specific C-reactive protein (hsCRP) blood levels | during the study conduct
To assess the tumor necrosing factor alpha (TNFα) blood levels | during the study conduct

SECONDARY OUTCOMES:
TEAEs collection | From the signature of the informed consent up to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Stan Glezer, Study Director — Sanofi